CLINICAL TRIAL: NCT01856309
Title: A Multicenter, Parallel-group Study of Long-term Safety and Efficacy of CNTO 136 (Sirukumab) for Rheumatoid Arthritis in Subjects Completing Treatment in Studies CNTO136ARA3002 (SIRROUND-D) and CNTO136ARA3003 (SIRROUND-T)
Brief Title: Long-term Safety and Efficacy of Sirukumab in Participants With RA Completing Studies CNTO136ARA3002 or CNTO136ARA3003
Acronym: SIRROUND-LTE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR102023; CNTO136ARA3004 (Other: Janssen Research & Development, LLC); 2012-001176-10 (EudraCT Number)
Record Dates: First submitted 2013-05-15; First posted 2013-05-17 (Estimated); Results first posted 2019-05-06 (Actual); Last update posted 2019-05-06 (Actual); Status verified 2019-04

CONDITIONS: Arthritis, Rheumatoid
Keywords: Rheumatoid Arthritis; Sirukumab; CNTO 136; CNTO136ARA3002; SIRROUND-D; CNTO136ARA3003; SIRROUND-T; SIRROUND-LTE
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — sirukumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sirukumab 100 mg (Experimental)
  Interventions: Drug: Sirukumab 100 mg
- Sirukumab 50 mg / placebo (Experimental)
  Interventions: Drug: Sirukumab 50 mg; Drug: Placebo

INTERVENTIONS:
Drug: Sirukumab 100 mg — Sirukumab 100 mg subcutaneously (SC) at Weeks 0 (administered as the last dose in CNTO136ARA3002 or CNTO136ARA3003), 2, and every 2 weeks through Week 156 for participants who completed CNTO136ARA3002 and through Week 208 for participants who completed CNTO136ARA3003.
  Arms: Sirukumab 100 mg
Drug: Sirukumab 50 mg — Sirukumab 50 mg SC at Weeks 0 (administered as the last dose in CNTO136ARA3002 or CNTO136ARA3003), 4, and every 4 weeks through Week 156 for participants who completed CNTO136ARA3002 and through Week 208 for participants who completed CNTO136ARA3003.
  Arms: Sirukumab 50 mg / placebo
Drug: Placebo — Between sirukumab 50 mg injections, placebo SC injections will be administered at Weeks 2, 6, and every 4 weeks until the study becomes open-label, and placebo injections are discontinued.
  Arms: Sirukumab 50 mg / placebo

SUMMARY:
The purpose of this study is to evaluate the long-term safety and efficacy of CNTO 136 (sirukumab) in participants with rheumatoid arthritis (RA) who are unresponsive to treatment with modifying antirheumatic drugs (DMARDs) or anti-TNF alpha agents.

DETAILED DESCRIPTION:
This is a multicenter, long-term study of sirukumab (CNTO 136) that will be conducted in two groups of participants at the same time (parallel-group study). The maximum duration of participation in this study is 208 weeks, followed by approximately 16 weeks of safety and efficacy follow-up after the administration of the final study agent injection of sirukumab. Participant safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Completed participation in Studies CNTO136ARA3002 or CNTO136ARA3003
* Signed an informed consent form (ICF) indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study
* Signed an informed consent form (ICF) for pharmacogenetics research (how a person's genes may affect a drug's effects) in order to participate in the optional pharmacogenetics component of this study. Refusal to give consent for this component does not exclude a participant from participation in this clinical study

Exclusion Criteria:

* Withdraws consent and/or discontinues participation in study CNTO136ARA3002 or CNTO136ARA3003
* Is pregnant
* Has active diverticulitis
* Has any condition that, in the opinion of the investigator, would make participation not be in the best interest (eg, compromise the well-being) of the participant or that could prevent, limit, or confound the protocol-specified assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1820 (Actual)
Dates: Start 2013-08-07 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (197):
- United States (66):
  - Birmingham, Alabama
  - Glendale, Arizona
  - Mesa, Arizona
  - Peoria, Arizona
  - Phoenix, Arizona
  - Covina, California
  - El Cajon, California
  - Glendale, California
  - Hemet, California
  - Huntington Beach, California
  - La Jolla, California
  - La Palma, California
  - Placentia, California
  - Upland, California
  - Victorville, California
  - Whittier, California
  - Hamden, Connecticut
  - Aventura, Florida
  - Boca Raton, Florida
  - Brandon, Florida
  - Daytona Beach, Florida
  - DeBary, Florida
  - Miami, Florida
  - Orlando, Florida
  - Palm Harbor, Florida
  - Plantation, Florida
  - Sarasota, Florida
  - Tampa, Florida
  - Zephyrhills, Florida
  - Cedar Rapids, Iowa
  - Bowling Green, Kentucky
  - Monroe, Louisiana
  - Cumberland, Maryland
  - Hagerstown, Maryland
  - Wheaton, Maryland
  - Rochester, Minnesota
  - Flowood, Mississippi
  - Springfield, Missouri
  - St Louis, Missouri
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Freehold, New Jersey
  - Albuquerque, New Mexico
  - Brooklyn, New York
  - Charlotte, North Carolina
  - Cincinnati, Ohio
  - Columbus, Ohio
  - Dayton, Ohio
  - Middleburg Heights, Ohio
  - Edmond, Oklahoma
  - Tulsa, Oklahoma
  - Duncansville, Pennsylvania
  - Wyomissing, Pennsylvania
  - Charleston, South Carolina
  - Austin, Texas
  - Carrollton, Texas
  - Corpus Christi, Texas
  - Cypress, Texas
  - Dallas, Texas
  - Houston, Texas
  - Katy, Texas
  - Lubbock, Texas
  - Mesquite, Texas
  - Victoria, Texas
  - Beckley, West Virginia
  - Clarksburg, West Virginia
- Argentina (3):
  - Buenos Aires
  - Rosario
  - San Miguel de Tucumán
- Victoria Park, Australia
- Vienna, Austria
- Liège, Belgium
- Bulgaria (2):
  - Plovdiv
  - Sofia
- Canada (3):
  - Victoria, British Columbia
  - Winnipeg, Manitoba
  - Edmonton
- Chile (3):
  - Rancagua
  - Santiago
  - Valdivia
- Colombia (3):
  - Bogotá
  - Chía
  - Medellín
- Croatia (3):
  - Osijek
  - Rijeka
  - Zagreb
- Toulouse, France
- Germany (7):
  - Berlin
  - Cologne
  - Frankfurt am Main
  - Göttingen
  - Hamburg
  - Vogelsang-Gommern
  - Würzburg
- Japan (37):
  - Ayauta
  - Bunkyō City
  - Fukuoka
  - Higashihiroshima
  - Hiroshima
  - Izumo
  - Kagoshima
  - Katō
  - Kawagoe
  - Kita-Gun
  - Kumamoto
  - Kurume
  - Matsuyama
  - Miyazaki
  - Nagano
  - Nagasaki
  - Nagoya
  - Nishimuro-gun
  - Nishinomiya
  - Okayama
  - Osaka
  - Sapporo
  - Sasebo
  - Shibata
  - Shimonoseki
  - Shimotsuke
  - Shinjuku-ku
  - Sumida-ku
  - Takaoka,Toyama
  - Takasaki
  - Tokorozawa
  - Tokushima
  - Tomishiro
  - Tonami
  - Tsu
  - Ureshino
  - Yokohama
- Lithuania (4):
  - Alytus
  - Kaunas
  - Klaipėda
  - Šiauliai
- Malaysia (2):
  - Kuala Lumpur
  - Kuching
- Mexico (7):
  - Cuernavaca
  - Guadalajara
  - Mexicali
  - Mérida
  - México
  - Morelia
  - San Luis de Potosi
- Sneek, Netherlands
- Poland (7):
  - Bialystok
  - Bydgoszcz
  - Elblag
  - Lublin
  - Poznan
  - Ustroń
  - Warsaw
- Lisbon, Portugal
- San Juan, Puerto Rico
- Romania (2):
  - Bucharest
  - Iași
- Russia (11):
  - Barnaul
  - Moscow
  - Novosibirsk
  - Omsk
  - Orenburg
  - Ryazan
  - Saint Petersburg
  - Saratov
  - Smolensk
  - Ulyanovsk
  - Yaroslavl
- Serbia (3):
  - Belgrade
  - Kragujevac
  - Niška Banja
- South Africa (3):
  - Cape Town
  - Port Elizabeth
  - Pretoria
- South Korea (10):
  - Busan
  - Daegu
  - Daejeon
  - Gwangju
  - Incheon
  - Jeonju
  - Namdong-Gu
  - Seongnam-si
  - Seoul
  - Suwon
- Spain (4):
  - A Coruña
  - Barakaldo
  - Santander
  - Santiago de Compostela
- Taiwan (3):
  - Kaohsiung City
  - Taichung
  - Taipei
- Ukraine (5):
  - Kharkiv
  - Kyiv
  - Odesa
  - Vinnytsia
  - Zaporizhzhia
- United Kingdom (2):
  - London
  - Wigan

REFERENCES:
- [Derived] Aletaha D, Bingham CO, Karpouzas GA, Takeuchi T, Thorne C, Bili A, Agarwal P, Hsu B, Rao R, Brown K, Tanaka Y. Long-term safety and efficacy of sirukumab for patients with rheumatoid arthritis who previously received sirukumab in randomised controlled trials (SIRROUND-LTE). RMD Open. 2021 Jan;7(1):e001465. doi: 10.1136/rmdopen-2020-001465. PMID 33526709

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who completed participation in studies CNTO136ARA3002 (NCT01604343) and CNTO136ARA3003 (NCT01606761) and consented to participate in extension study were enrolled in this study.
Pre-assignment Details: Data in the participant flow section is reported for treatment discontinuation.
Groups:
- Placebo to 50 mg q4w Due to EE/LE/CO: Participants initially randomized to placebo, then at early escape (EE), late escape (LE), or cross over (CO) randomized to sirukumab 50 milligram (mg) every 4 weeks (q4w) during the primary studies CNTO136ARA3002 and CNTO136ARA3003, and then continued to receive the same regimen (sirukumab 50 mg q4w) upon entering this long-term extension (LTE) study.
- Placebo to 100 mg q2w Due to EE/LE/CO: Participants initially randomized to placebo, then at EE, LE, or CO randomized to sirukumab 100 mg every two weeks (q2w) during the primary studies CNTO136ARA3002 and CNTO136ARA3003, and then continued to receive the same regimen upon entering this LTE study.
- Sirukumab 50 mg q4w: Participants initially randomized to sirukumab 50 mg q4w during the primary studies CNTO136ARA3002 and CNTO136ARA3003, and then continued to receive the same regimen upon entering this LTE study.
- Sirukumab 100 mg q2w: Participants initially randomized to sirukumab 100 mg q2w during the primary studies CNTO136ARA3002 and CNTO136ARA3003, and then continued to receive the same regimen upon entering this LTE study.
Period: Overall Study
Arm/Group | Placebo to 50 mg q4w Due to EE/LE/CO | Placebo to 100 mg q2w Due to EE/LE/CO | Sirukumab 50 mg q4w | Sirukumab 100 mg q2w
Started | 305 | 291 | 606 | 618
Participants From Study CNTO136ARA3002 | 197 | 187 | 405 | 412
Participants From Study CNTO136ARA3003 | 108 | 104 | 201 | 206
Treated Partcipants | 305 | 290 | 605 | 618
Completed | 6 | 3 | 11 | 9
Not Completed | 299 | 288 | 595 | 609
Not completed — Death | 4 | 6 | 11 | 6
Not completed — Lost to Follow-up | 6 | 2 | 4 | 8
Not completed — Withdrawal by Subject | 11 | 13 | 28 | 26
Not completed — Other | 227 | 225 | 447 | 469
Not completed — Lack of Efficacy | 14 | 9 | 40 | 25
Not completed — Adverse Event | 31 | 31 | 55 | 65
Not completed — Pregnancy | 0 | 0 | 0 | 1
Not completed — Physician Decision | 6 | 1 | 6 | 8
Not completed — Noncompliance With Study Drug | 0 | 1 | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Placebo to 50 mg q4w Due to EE/LE/CO: Participants initially randomized to placebo, then at early escape (EE), late escape (LE), or cross over (CO) randomized to sirukumab 50 mg every 4 weeks (q4w) during the primary studies CNTO136ARA3002 and CNTO136ARA3003, and then continued to receive the same regimen (sirukumab 50 mg q4w) upon entering this long-term extension (LTE) study.
- Total: Total of all reporting groups
Arm/Group | Placebo to 50 mg q4w Due to EE/LE/CO | Placebo to 100 mg q2w Due to EE/LE/CO | Sirukumab 50 mg q4w | Sirukumab 100 mg q2w | Total
Number analyzed (Participants) | 305 | 291 | 606 | 618 | 1820
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (11.92) | 53.1 (11.75) | 53.1 (11.43) | 53.4 (11.29) | 53.4 (11.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 241 | 231 | 479 | 503 | 1454
  Male | 64 | 60 | 127 | 115 | 366
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3 | 5 | 11
  Asian | 50 | 47 | 102 | 110 | 309
  Black or African American | 10 | 15 | 21 | 23 | 69
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  White | 231 | 211 | 433 | 443 | 1318
  Other | 11 | 15 | 40 | 31 | 97
  Multiple | 0 | 0 | 0 | 1 | 1
  Not reported | 1 | 2 | 5 | 4 | 12
  Unknown | 0 | 0 | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 4 | 5 | 4 | 2 | 15
  Australia | 0 | 1 | 1 | 0 | 2
  Austria | 1 | 1 | 0 | 0 | 2
  Belgium | 0 | 1 | 0 | 0 | 1
  Bulgaria | 0 | 3 | 3 | 3 | 9
  Canada | 2 | 0 | 2 | 3 | 7
  Chile | 11 | 7 | 14 | 18 | 50
  Colombia | 2 | 6 | 10 | 11 | 29
  Croatia | 1 | 2 | 3 | 2 | 8
  France | 0 | 0 | 1 | 0 | 1
  Germany | 2 | 3 | 10 | 5 | 20
  Italy | 1 | 0 | 0 | 1 | 2
  Japan | 36 | 36 | 74 | 78 | 224
  Lithuania | 13 | 10 | 26 | 32 | 81
  Malaysia | 3 | 0 | 1 | 1 | 5
  Mexico | 17 | 16 | 39 | 40 | 112
  Netherlands | 1 | 2 | 1 | 1 | 5
  Poland | 36 | 31 | 67 | 62 | 196
  Portugal | 3 | 0 | 3 | 4 | 10
  Puerto Rico | 1 | 0 | 3 | 0 | 4
  Romania | 2 | 0 | 2 | 4 | 8
  Russia | 34 | 29 | 63 | 72 | 198
  Serbia | 21 | 23 | 38 | 36 | 118
  South Africa | 13 | 16 | 22 | 20 | 71
  Korea, Republic Of | 6 | 5 | 14 | 23 | 48
  Spain | 3 | 2 | 5 | 4 | 14
  Taiwan, Province Of China | 5 | 6 | 12 | 4 | 27
  Ukraine | 16 | 13 | 31 | 41 | 101
  United Kingdom | 0 | 0 | 1 | 2 | 3
  United States | 71 | 73 | 156 | 149 | 449

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Serious Adverse Events (SAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: From baseline of this LTE study up to 4.3 years
Population: Population included all participants who were enrolled in this study. One participant who mistakenly took sirukumab 100mg, when was originally assigned to sirukumab 50mg, was analyzed under the sirukumab 100mg group for all safety analyses.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo to 50 mg q4w Due to EE/LE/CO | Placebo to 100 mg q2w Due to EE/LE/CO | Sirukumab 50 mg q4w | Sirukumab 100 mg q2w
Number analyzed (Participants) | 305 | 291 | 605 | 619
Percentage of participants | 21.3 | 27.8 | 26.4 | 23.1

2. Primary Outcome: Percentage of Participants With Major Adverse Cardiovascular Events (MACE)
Description: MACE was defined as a composite of Myocardial Infarction (MI), stroke, death, hospitalization for unstable angina, and hospitalization for Transient Ischemic Attack (TIA). Adjudication of these events by the Endpoint Adjudication Committee (EAC) was performed in a blinded fashion.
Time Frame: From baseline of this LTE study up to 4.3 years
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo to 50 mg q4w Due to EE/LE/CO | Placebo to 100 mg q2w Due to EE/LE/CO | Sirukumab 50 mg q4w | Sirukumab 100 mg q2w
Number analyzed (Participants) | 305 | 291 | 605 | 619
Percentage of participants | 2.0 | 0.7 | 2.3 | 1.1

3. Primary Outcome: Percentage of Participants With Malignancies
Description: Percentage of participants with one or more malignancy was reported.
Time Frame: From baseline of this LTE study up to 4.3 years
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo to 50 mg q4w Due to EE/LE/CO | Placebo to 100 mg q2w Due to EE/LE/CO | Sirukumab 50 mg q4w | Sirukumab 100 mg q2w
Number analyzed (Participants) | 305 | 291 | 605 | 619
Percentage of participants | 1.0 | 3.4 | 1.5 | 1.8

4. Primary Outcome: Percentage of Participants With Serious Infections
Description: Percentage of participants with one or more serious infections was reported.
Time Frame: From baseline of this LTE study up to 4.3 years
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo to 50 mg q4w Due to EE/LE/CO | Placebo to 100 mg q2w Due to EE/LE/CO | Sirukumab 50 mg q4w | Sirukumab 100 mg q2w
Number analyzed (Participants) | 305 | 291 | 605 | 619
Percentage of participants | 7.9 | 12.0 | 10.4 | 10.7

5. Primary Outcome: Percentage of Participants With Gastrointestinal (GI) Perforations
Description: Percentage of participants with one or more GI perforations was reported. GI perforation is a hole that develops through the entire wall of the stomach, small intestine, large bowel, or gallbladder.
Time Frame: From baseline of this LTE study up to 4.3 years
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo to 50 mg q4w Due to EE/LE/CO | Placebo to 100 mg q2w Due to EE/LE/CO | Sirukumab 50 mg q4w | Sirukumab 100 mg q2w
Number analyzed (Participants) | 305 | 291 | 605 | 619
Percentage of participants | 0.7 | 1.4 | 0.7 | 0.5

6. Primary Outcome: Percentage of Participants With Hepatobiliary Abnormalities
Description: Percentage of participants with hepatobiliary abnormalities was reported.
Time Frame: From baseline of this LTE study up to 4.3 years
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo to 50 mg q4w Due to EE/LE/CO | Placebo to 100 mg q2w Due to EE/LE/CO | Sirukumab 50 mg q4w | Sirukumab 100 mg q2w
Number analyzed (Participants) | 305 | 291 | 605 | 619
Percentage of participants | 0 | 0.3 | 0.2 | 0.2

7. Primary Outcome: Percentage of Participants With Serious or Moderate/Severe Systemic Hypersensitivity Reactions, or Serum Sickness Adverse Events
Description: Percentage of participants with serious or moderate/severe systemic hypersensitivity reactions, or serum sickness adverse events (AEs) was reported.
Time Frame: From baseline of this LTE study up to 4.3 years
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo to 50 mg q4w Due to EE/LE/CO | Placebo to 100 mg q2w Due to EE/LE/CO | Sirukumab 50 mg q4w | Sirukumab 100 mg q2w
Number analyzed (Participants) | 305 | 291 | 605 | 619
Percentage of participants | 0.3 | 0.7 | 0.2 | 0.3

8. Secondary Outcome: Percentage of Participants With Toxicity Grade 4 Decrease in Neutrophils
Description: Percentage of participants with toxicity grade 4 decrease in neutrophils was reported. As per National Cancer Institute's Common Terminology Criteria for Adverse Events, toxicity grade 4 was defined as decrease in neutrophils less than (<) 500 per Cubic Millimeter (mm^3) or < 0.5 * 10^9 per liter.
Time Frame: From baseline of primary studies through end of this LTE study (Approximately 5.3 years)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo to 50 mg q4w Due to EE/LE/CO | Placebo to 100 mg q2w Due to EE/LE/CO | Sirukumab 50 mg q4w | Sirukumab 100 mg q2w
Number analyzed (Participants) | 305 | 291 | 605 | 619
Percentage of participants | 1.3 | 0 | 0.5 | 0

9. Secondary Outcome: Percentage of Participants With Toxicity Grade 4 Decrease in Platelets
Description: Percentage of participants with toxicity grade 4 decrease in platelets was reported. As per National Cancer Institute's Common Terminology Criteria for Adverse Events, toxicity grade 4 was defined as decreased in platelets <25000/mm^3 or < 25.0 * 10^9 per liter.
Time Frame: From baseline of primary studies through end of this LTE study (Approximately 5.3 years)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo to 50 mg q4w Due to EE/LE/CO | Placebo to 100 mg q2w Due to EE/LE/CO | Sirukumab 50 mg q4w | Sirukumab 100 mg q2w
Number analyzed (Participants) | 305 | 291 | 605 | 619
Percentage of participants | 0 | 0 | 0 | 0

10. Secondary Outcome: Percentage of Participants With ALT >= 3*ULN, ALT >= 5*ULN and ALT >= 8*ULN
Description: Percentage of participants with Alanine Aminotranserase (ALT) >= 3*Upper Limit of Normal (ULN), ALT >= 5*ULN or ALT >= 8*ULN was reported.
Time Frame: From baseline of primary studies through end of this LTE study (Approximately 5.3 years)
Population: Population included all participants who were enrolled in this study. 1 participant who mistakenly took sirukumab 100mg, when was originally assigned to sirukumab 50mg, was analyzed under the sirukumab 100mg group for all safety analyses.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo to 50 mg q4w Due to EE/LE/CO | Placebo to 100 mg q2w Due to EE/LE/CO | Sirukumab 50 mg q4w | Sirukumab 100 mg q2w
Number analyzed (Participants) | 305 | 291 | 605 | 619
Percentage of participants
  ALT >= 3 * ULN | 14.1 | 14.4 | 15.9 | 17.1
  ALT >= 5 * ULN | 2.0 | 2.4 | 2.5 | 3.9
  ALT >= 8 * ULN | 0 | 0.7 | 0.2 | 0.2

11. Secondary Outcome: Percentage of Participants With AST >= 3*ULN, AST >= 5*ULN and AST >= 8*ULN
Description: Percentage of participants with Aspartate Aminotransferase (AST) >= 3*ULN, AST >= 5*ULN and AST >= 8*ULN was reported.
Time Frame: From baseline of primary studies through end of this LTE study (Approximately 5.3 years)
Population: as for outcome 10
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo to 50 mg q4w Due to EE/LE/CO | Placebo to 100 mg q2w Due to EE/LE/CO | Sirukumab 50 mg q4w | Sirukumab 100 mg q2w
Number analyzed (Participants) | 305 | 291 | 605 | 619
Percentage of participants
  AST >= 3 * ULN | 3.9 | 6.2 | 4.5 | 7.8
  AST >= 5 * ULN | 0.3 | 1.7 | 0.5 | 1.1
  AST >= 8 * ULN | 0 | 0 | 0 | 0.3

12. Secondary Outcome: Percentage of Participants With Either ALT >= 3*ULN or AST >= 3*ULN, and Total Bilirubin >= 2*ULN
Description: Percentage of participants with either ALT >= 3*ULN or AST >= 3*ULN and total bilirubin >= 2*ULN was reported.
Time Frame: From baseline of primary studies through end of this LTE study (Approximately 5.3 years)
Population: as for outcome 10
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo to 50 mg q4w Due to EE/LE/CO | Placebo to 100 mg q2w Due to EE/LE/CO | Sirukumab 50 mg q4w | Sirukumab 100 mg q2w
Number analyzed (Participants) | 305 | 291 | 605 | 619
Percentage of participants | 0 | 0 | 0 | 0.2

13. Secondary Outcome: Percentage of Participants With Normal Total Cholesterol Value at Baseline and at Least 1 Abnormal Value Post-Baseline
Description: Percentage of participants with normal total cholesterol value at baseline and at least 1 abnormal value post-baseline was reported. Abnormal total cholesterol value was defined as total cholesterol value more than (>) 200 milligrams per deciliter (mg/dL).
Time Frame: From baseline of primary studies through end of this LTE study (Approximately 5.3 years)
Population: Population included all participants who were enrolled in this study and had total cholesterol baseline value within normal range.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo to 50 mg q4w Due to EE/LE/CO | Placebo to 100 mg q2w Due to EE/LE/CO | Sirukumab 50 mg q4w | Sirukumab 100 mg q2w
Number analyzed (Participants) | 177 | 163 | 354 | 345
Percentage of participants | 86.4 | 81.6 | 82.5 | 87.2

14. Secondary Outcome: Percentage of Participants With Normal Low-Density Lipoprotein (LDL) Value at Baseline and at Least 1 Abnormal Value Post-Baseline
Description: Percentage of participants with normal LDL value at baseline and at least 1 abnormal value post-baseline was reported. Abnormal LDL value was defined as LDL value > 130 mg/dL.
Time Frame: From baseline of primary studies through end of this LTE study (Approximately 5.3 years)
Population: Population included all participants who were enrolled in this study and had LDL baseline value within normal range.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo to 50 mg q4w Due to EE/LE/CO | Placebo to 100 mg q2w Due to EE/LE/CO | Sirukumab 50 mg q4w | Sirukumab 100 mg q2w
Number analyzed (Participants) | 225 | 209 | 459 | 449
Percentage of participants | 70.2 | 67.9 | 69.7 | 70.8

15. Secondary Outcome: Percentage of Participants With Normal High-Density Lipoprotein (HDL) Value at Baseline and at Least 1 Abnormal Value Post-Baseline
Description: Percentage of participants with normal HDL value at baseline and at least 1 abnormal value post-baseline was reported. Abnormal HDL value was defined as HDL value < 40 mg/dL.
Time Frame: From baseline of primary studies through end of this LTE study (Approximately 5.3 years)
Population: Population included all participants who were enrolled in this study and had HDL baseline value within normal range.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo to 50 mg q4w Due to EE/LE/CO | Placebo to 100 mg q2w Due to EE/LE/CO | Sirukumab 50 mg q4w | Sirukumab 100 mg q2w
Number analyzed (Participants) | 277 | 273 | 533 | 569
Percentage of participants | 16.2 | 14.7 | 16.1 | 16.0

16. Secondary Outcome: Percentage of Participants With Normal Triglyceride Value at Baseline and at Least 1 Abnormal Value Post-Baseline
Description: Percentage of participants with normal triglyceride value at baseline and at least 1 abnormal value post-baseline was reported. Abnormal triglyceride value was defined as triglyceride value > 250 mg/dL.
Time Frame: From baseline of primary studies through end of this LTE study (Approximately 5.3 years)
Population: Population included all participants who were enrolled in this study and had triglyceride baseline value within normal range.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo to 50 mg q4w Due to EE/LE/CO | Placebo to 100 mg q2w Due to EE/LE/CO | Sirukumab 50 mg q4w | Sirukumab 100 mg q2w
Number analyzed (Participants) | 279 | 268 | 554 | 564
Percentage of participants | 32.6 | 35.1 | 36.1 | 34.4

17. Secondary Outcome: Percentage of Participants Who Achieved American College of Rheumatology (ACR) 50 Response Through Week 260
Description: ACR 50 response is greater than or equal to (>=) 50 percent (%) improvement in both tender joint count (68) and swollen joint count (66) and >= 50% improvement in 3 of following 5 assessments:Participant's assessment of pain using visual analog scale (VAS) (0-10 scale, 0=no pain and 10=worst possible pain),Participant's global assessment of disease activity by using VAS (scale ranges from 0 to 10, [0 = very well to 10 = very poor]), Physician's global assessment of disease activity using VAS (scale ranges from 0 to 10, [0=no arthritis activity to 10=extremely active arthritis]), Participant's assessment of physical function as measured by Health Assessment Questionnaire-Disability Index (HAQ-DI) (scale ranges from 0= no difficulty to 3= inability to perform a task in that area), and Serum C-reactive protein (CRP). Participants were analyzed for efficacy according to assigned treatment groups from the primary studies, regardless of treatments actually received.
Time Frame: Week 2, 4, 6, 8, 12, 16, 18, 20, 24, 28, 32, 36, 40, 44, 48, 52, 76, 80, 104, 128, 132, 156, 180, 208, 232 and 260
Population: Population included all participants who were enrolled in this study. For "Placebo to 50mg" and "Placebo to 100mg" groups, only efficacy data collected after escape or CO (after Week 18) to sirukumab was planned to be reported, with exception of baseline data. Here 'n' signifies the number of participants analyzed at the specified time point.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo to 50 mg q4w Due to EE/LE/CO | Placebo to 100 mg q2w Due to EE/LE/CO | Sirukumab 50 mg q4w | Sirukumab 100 mg q2w
Number analyzed (Participants) | 305 | 291 | 606 | 618
Percentage of participants
  At Week 2: number analyzed (Participants) | 0 | 0 | 604 | 615
  At Week 2 |  |  | 2.5 | 2.4
  At Week 4: number analyzed (Participants) | 0 | 0 | 603 | 614
  At Week 4 |  |  | 9.1 | 9.7
  At Week 6: number analyzed (Participants) | 0 | 0 | 511 | 527
  At Week 6 |  |  | 16.2 | 14.6
  At Week 8: number analyzed (Participants) | 0 | 0 | 603 | 611
  At Week 8 |  |  | 21.4 | 20.0
  At Week 12: number analyzed (Participants) | 0 | 0 | 600 | 614
  At Week 12 |  |  | 27.7 | 29.6
  At Week 16: number analyzed (Participants) | 0 | 0 | 603 | 614
  At Week 16 |  |  | 31.8 | 29.2
  At Week 18: number analyzed (Participants) | 0 | 0 | 602 | 612
  At Week 18 |  |  | 33.7 | 32.0
  At Week 20: number analyzed (Participants) | 111 | 106 | 602 | 611
  At Week 20 | 4.5 | 3.8 | 36.9 | 38.1
  At Week 24: number analyzed (Participants) | 112 | 106 | 606 | 615
  At Week 24 | 17.9 | 10.4 | 35.1 | 37.9
  At Week 28: number analyzed (Participants) | 180 | 173 | 600 | 612
  At Week 28 | 24.4 | 23.1 | 40.0 | 39.2
  At Week 32: number analyzed (Participants) | 180 | 169 | 602 | 614
  At Week 32 | 30.0 | 30.2 | 40.9 | 42.2
  At Week 36: number analyzed (Participants) | 178 | 174 | 601 | 612
  At Week 36 | 29.2 | 33.9 | 42.3 | 43.0
  At Week 40: number analyzed (Participants) | 175 | 173 | 595 | 612
  At Week 40 | 38.3 | 34.7 | 42.0 | 42.2
  At Week 44: number analyzed (Participants) | 187 | 179 | 598 | 609
  At Week 44 | 40.1 | 33.5 | 43.3 | 44.3
  At Week 48: number analyzed (Participants) | 187 | 179 | 601 | 608
  At Week 48 | 43.3 | 27.9 | 44.6 | 44.1
  At Week 52: number analyzed (Participants) | 191 | 182 | 605 | 617
  At Week 52 | 41.9 | 34.1 | 43.0 | 44.9
  At Week 76: number analyzed (Participants) | 196 | 185 | 401 | 410
  At Week 76 | 56.6 | 49.7 | 52.4 | 56.1
  At Week 80: number analyzed (Participants) | 90 | 87 | 178 | 187
  At Week 80 | 38.9 | 26.4 | 38.2 | 44.9
  At Week 104: number analyzed (Participants) | 283 | 267 | 571 | 575
  At Week 104 | 48.8 | 46.1 | 50.3 | 53.0
  At Week 128: number analyzed (Participants) | 76 | 73 | 157 | 157
  At Week 128 | 35.5 | 43.8 | 42.7 | 46.5
  At Week 132: number analyzed (Participants) | 174 | 165 | 356 | 369
  At Week 132 | 51.1 | 46.7 | 50.0 | 53.4
  At Week 156: number analyzed (Participants) | 242 | 227 | 499 | 506
  At Week 156 | 48.3 | 56.4 | 50.3 | 52.6
  At Week 180: number analyzed (Participants) | 184 | 175 | 381 | 390
  At Week 180 | 53.3 | 54.9 | 54.6 | 56.4
  At Week 208: number analyzed (Participants) | 110 | 93 | 199 | 213
  At Week 208 | 50.9 | 50.5 | 50.8 | 59.6
  At Week 232: number analyzed (Participants) | 33 | 28 | 66 | 70
  At Week 232 | 48.5 | 57.1 | 51.5 | 57.1
  At Week 260: number analyzed (Participants) | 3 | 2 | 10 | 4
  At Week 260 | 66.7 | 50.0 | 60.0 | 25.0

18. Secondary Outcome: Percentage of Participants With Boolean-Based American College of Rheumatology (ACR) or European League Against Rheumatism (EULAR) Remission Through Week 260
Description: Boolean based ACR/EULAR remission is achieved if all of the following 4 criteria at that visit are met: tender joint count (68 joints) <=1; swollen joint count (66 joints) <=1; CRP <=1 milligram per deciliter (mg/dL); and patient's global assessment of disease activity on visual analog scale (VAS) <=1 on a 0 (very well ) to 10 (extremely bad) scale. Higher scores indicates worst health condition. Participants were analyzed for efficacy according to the assigned treatment groups from the primary studies, regardless of the treatments they actually received.
Time Frame: Week 2, 4, 6, 8, 12, 16, 18, 20, 24, 28, 32, 36, 40, 44, 48, 52, 76, 80, 104, 128, 132, 156, 180, 208, 232 and 260
Population: as for outcome 17
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo to 50 mg q4w Due to EE/LE/CO | Placebo to 100 mg q2w Due to EE/LE/CO | Sirukumab 50 mg q4w | Sirukumab 100 mg q2w
Number analyzed (Participants) | 305 | 291 | 606 | 618
Percentage of participants
  At Week 2: number analyzed (Participants) | 0 | 0 | 604 | 616
  At Week 2 |  |  | 0.2 | 0.2
  At Week 4: number analyzed (Participants) | 0 | 0 | 603 | 616
  At Week 4 |  |  | 0.5 | 0.6
  At Week 6: number analyzed (Participants) | 0 | 0 | 511 | 527
  At Week 6 |  |  | 0.8 | 1.5
  At Week 8: number analyzed (Participants) | 0 | 0 | 603 | 611
  At Week 8 |  |  | 1.2 | 2.5
  At Week 12: number analyzed (Participants) | 0 | 0 | 602 | 614
  At Week 12 |  |  | 3.2 | 4.9
  At Week 16: number analyzed (Participants) | 0 | 0 | 603 | 614
  At Week 16 |  |  | 3.3 | 5.7
  At Week 18: number analyzed (Participants) | 0 | 0 | 603 | 613
  At Week 18 |  |  | 4.3 | 5.4
  At Week 20: number analyzed (Participants) | 111 | 106 | 604 | 611
  At Week 20 | 0 | 0 | 4.5 | 5.9
  At Week 24: number analyzed (Participants) | 112 | 106 | 606 | 615
  At Week 24 | 0.9 | 0.9 | 5.3 | 8.1
  At Week 28: number analyzed (Participants) | 180 | 174 | 602 | 613
  At Week 28 | 2.8 | 2.9 | 6.0 | 6.2
  At Week 32: number analyzed (Participants) | 180 | 170 | 601 | 613
  At Week 32 | 2.2 | 4.1 | 4.8 | 7.7
  At Week 36: number analyzed (Participants) | 178 | 174 | 603 | 611
  At Week 36 | 2.8 | 4.0 | 7.8 | 9.7
  At Week 40: number analyzed (Participants) | 177 | 173 | 596 | 613
  At Week 40 | 4.0 | 6.4 | 7.2 | 9.0
  At Week 44: number analyzed (Participants) | 187 | 180 | 598 | 610
  At Week 44 | 4.3 | 6.1 | 7.4 | 9.7
  At Week 48: number analyzed (Participants) | 187 | 179 | 602 | 609
  At Week 48 | 4.3 | 7.3 | 9.8 | 9.0
  At Week 52: number analyzed (Participants) | 190 | 181 | 604 | 618
  At Week 52 | 6.8 | 6.6 | 9.3 | 7.1
  At Week 76: number analyzed (Participants) | 196 | 183 | 402 | 411
  At Week 76 | 9.7 | 7.1 | 10.7 | 9.2
  At Week 80: number analyzed (Participants) | 91 | 87 | 180 | 189
  At Week 80 | 6.6 | 8.0 | 7.8 | 6.3
  At Week 104: number analyzed (Participants) | 283 | 270 | 573 | 578
  At Week 104 | 10.6 | 11.1 | 12.6 | 10.2
  At Week 128: number analyzed (Participants) | 76 | 74 | 158 | 157
  At Week 128 | 2.6 | 8.1 | 10.8 | 8.9
  At Week 132: number analyzed (Participants) | 177 | 168 | 360 | 373
  At Week 132 | 12.4 | 11.3 | 10.8 | 10.2
  At Week 156: number analyzed (Participants) | 244 | 229 | 503 | 508
  At Week 156 | 9.4 | 8.7 | 10.9 | 11.8
  At Week 180: number analyzed (Participants) | 187 | 177 | 386 | 395
  At Week 180 | 11.8 | 10.7 | 14.2 | 13.9
  At Week 208: number analyzed (Participants) | 111 | 95 | 201 | 219
  At Week 208 | 12.6 | 13.7 | 11.4 | 19.2
  At Week 232: number analyzed (Participants) | 34 | 28 | 66 | 66
  At Week 232 | 11.8 | 17.9 | 18.2 | 9.1
  At Week 260: number analyzed (Participants) | 4 | 2 | 11 | 5
  At Week 260 | 0 | 0 | 18.2 | 0

19. Secondary Outcome: Percentage of Participants With Disease Activity Index Score 28 (CRP) Remission Through Week 260
Description: The Disease Activity Index Score 28 (DAS28) based on C-Reactive Protein (CRP) is a statistically derived index combining tender joints (28 joints), swollen joints (28 joints), CRP and patient's global assessment of disease activity. The set of 28 joint count is based on evaluation of the shoulder, elbow, wrist, metacarpophalangeal (MCP) MCP1 to MCP5, proximal interphalangeal (PIP) PIP1 to PIP5 joints of both the upper right extremity and the upper left extremity as well as the knee joints of lower right and lower left extremities. The values are 0=best to 10=worst. DAS28 (CRP) remission is defined as a DAS28 (CRP) value of less than (<) 2.6 at any study visit. Participants were analyzed for efficacy according to the assigned treatment groups from the primary studies, regardless of the treatments they actually received.
Time Frame: Week 2, 4, 6, 8, 12, 16, 18, 20, 24, 28, 32, 36, 40, 44, 48, 52, 76, 80, 104, 128, 132, 156, 180, 208, 232 and 260
Population: as for outcome 17
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo to 50 mg q4w Due to EE/LE/CO | Placebo to 100 mg q2w Due to EE/LE/CO | Sirukumab 50 mg q4w | Sirukumab 100 mg q2w
Number analyzed (Participants) | 305 | 291 | 606 | 618
Percentage of participants
  At Week 2: number analyzed (Participants) | 0 | 0 | 601 | 609
  At Week 2 |  |  | 2.7 | 2.6
  At Week 4: number analyzed (Participants) | 0 | 0 | 599 | 611
  At Week 4 |  |  | 7.5 | 9.0
  At Week 6: number analyzed (Participants) | 0 | 0 | 502 | 524
  At Week 6 |  |  | 10.2 | 13.4
  At Week 8: number analyzed (Participants) | 0 | 0 | 601 | 608
  At Week 8 |  |  | 15.0 | 18.8
  At Week 12: number analyzed (Participants) | 0 | 0 | 598 | 614
  At Week 12 |  |  | 20.4 | 23.5
  At Week 16: number analyzed (Participants) | 0 | 0 | 602 | 612
  At Week 16 |  |  | 23.8 | 24.0
  At Week 18: number analyzed (Participants) | 0 | 0 | 589 | 606
  At Week 18 |  |  | 25.6 | 25.4
  At Week 20: number analyzed (Participants) | 110 | 106 | 600 | 605
  At Week 20 | 1.8 | 0 | 29.8 | 30.1
  At Week 24: number analyzed (Participants) | 111 | 106 | 603 | 610
  At Week 24 | 7.2 | 7.5 | 30.8 | 32.1
  At Week 28: number analyzed (Participants) | 180 | 173 | 595 | 608
  At Week 28 | 17.8 | 20.8 | 33.8 | 32.7
  At Week 32: number analyzed (Participants) | 177 | 170 | 597 | 609
  At Week 32 | 24.9 | 24.7 | 35.3 | 36.9
  At Week 36: number analyzed (Participants) | 178 | 174 | 596 | 610
  At Week 36 | 21.3 | 30.5 | 35.1 | 35.4
  At Week 40: number analyzed (Participants) | 174 | 172 | 594 | 608
  At Week 40 | 29.9 | 32.0 | 34.5 | 34.9
  At Week 44: number analyzed (Participants) | 184 | 178 | 595 | 607
  At Week 44 | 34.2 | 30.9 | 36.0 | 35.4
  At Week 48: number analyzed (Participants) | 184 | 179 | 592 | 605
  At Week 48 | 33.2 | 31.3 | 38.7 | 38.3
  At Week 52: number analyzed (Participants) | 189 | 181 | 601 | 610
  At Week 52 | 30.7 | 32.6 | 38.8 | 37.4
  At Week 76: number analyzed (Participants) | 195 | 183 | 399 | 408
  At Week 76 | 44.6 | 44.3 | 47.6 | 45.8
  At Week 80: number analyzed (Participants) | 90 | 84 | 175 | 184
  At Week 80 | 38.9 | 39.3 | 38.3 | 38.6
  At Week 104: number analyzed (Participants) | 279 | 266 | 571 | 573
  At Week 104 | 44.8 | 47.4 | 42.6 | 46.6
  At Week 128: number analyzed (Participants) | 73 | 72 | 156 | 154
  At Week 128 | 43.8 | 43.1 | 45.5 | 43.5
  At Week 132: number analyzed (Participants) | 169 | 165 | 350 | 365
  At Week 132 | 41.4 | 47.3 | 48.0 | 49.0
  At Week 156: number analyzed (Participants) | 235 | 233 | 486 | 500
  At Week 156 | 43.0 | 47.1 | 46.5 | 49.6
  At Week 180: number analyzed (Participants) | 180 | 170 | 376 | 388
  At Week 180 | 48.9 | 48.8 | 50.5 | 53.9
  At Week 208: number analyzed (Participants) | 109 | 93 | 197 | 213
  At Week 208 | 55.0 | 54.8 | 54.3 | 60.1
  At Week 232: number analyzed (Participants) | 27 | 25 | 56 | 57
  At Week 232 | 59.3 | 52.0 | 57.1 | 59.6
  At Week 260: number analyzed (Participants) | 3 | 2 | 9 | 4
  At Week 260 | 66.7 | 100.0 | 77.8 | 25.0

20. Secondary Outcome: Change From Baseline in Clinical Disease Activity Index (CDAI) Score Through Week 260
Description: The CDAI score is a derived score of 4 components: tender joints (28 joints), swollen joints (28 joints), patient's global assessment of disease activity, and physician's global assessments of disease activity. The total score ranges from 0 to 76 with a lower score indicating less disease activity. A negative change in CDAI score indicates an improvement in disease activity and a positive change in score indicates a worsening of disease activity. Participants were analyzed for efficacy according to the assigned treatment groups from the primary studies, regardless of the treatments they actually received.
Time Frame: Baseline (Week 0 of primary studies), Week 2, 4, 6, 8, 12, 16, 18, 20, 24, 28, 32, 36, 40, 44, 48, 52, 76, 80, 104, 128, 132, 156, 180, 208, 232 and 260
Population: Population included all participants who were enrolled in this study. For "Placebo to 50mg" and "Placebo to 100mg" groups, only efficacy data collected after escape or CO (after Week 18) to sirukumab was planned to be reported, with exception of baseline data. Here 'n' signifies the number of participants analyzed at specified time point.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo to 50 mg q4w Due to EE/LE/CO | Placebo to 100 mg q2w Due to EE/LE/CO | Sirukumab 50 mg q4w | Sirukumab 100 mg q2w
Number analyzed (Participants) | 305 | 291 | 606 | 618
Units on a scale
  Change at Week 2: number analyzed (Participants) | 0 | 0 | 602 | 614
  Change at Week 2 |  |  | -6.54 (9.464) | -6.10 (9.295)
  Change at Week 4: number analyzed (Participants) | 0 | 0 | 598 | 614
  Change at Week 4 |  |  | -11.09 (11.257) | -10.73 (11.469)
  Change at Week 6: number analyzed (Participants) | 0 | 0 | 510 | 524
  Change at Week 6 |  |  | -13.79 (12.198) | -14.05 (11.613)
  Change at Week 8: number analyzed (Participants) | 0 | 0 | 602 | 611
  Change at Week 8 |  |  | -15.56 (12.736) | -15.74 (12.333)
  Change at Week 12: number analyzed (Participants) | 0 | 0 | 600 | 612
  Change at Week 12 |  |  | -17.79 (13.955) | -17.89 (13.636)
  Change at Week 16: number analyzed (Participants) | 0 | 0 | 600 | 612
  Change at Week 16 |  |  | -18.50 (13.956) | -18.65 (13.584)
  Change at Week 18: number analyzed (Participants) | 0 | 0 | 599 | 613
  Change at Week 18 |  |  | -18.93 (14.459) | -18.40 (13.524)
  Change at Week 20: number analyzed (Participants) | 109 | 106 | 601 | 610
  Change at Week 20 | -7.19 (12.051) | -7.01 (11.666) | -20.72 (14.077) | -19.96 (13.678)
  Change at Week 24: number analyzed (Participants) | 111 | 106 | 605 | 615
  Change at Week 24 | -15.08 (11.697) | -12.78 (11.654) | -21.20 (13.625) | -21.06 (13.888)
  Change at Week 28: number analyzed (Participants) | 179 | 172 | 600 | 612
  Change at Week 28 | -19.69 (13.518) | -19.58 (12.578) | -21.85 (14.000) | -21.33 (13.655)
  Change at Week 32: number analyzed (Participants) | 179 | 169 | 600 | 612
  Change at Week 32 | -20.36 (14.238) | -20.69 (12.754) | -22.37 (13.935) | -22.17 (13.462)
  Change at Week 36: number analyzed (Participants) | 177 | 174 | 600 | 611
  Change at Week 36 | -21.49 (12.343) | -22.53 (12.609) | -22.64 (13.750) | -22.79 (13.220)
  Change at Week 40: number analyzed (Participants) | 176 | 173 | 593 | 609
  Change at Week 40 | -22.67 (13.374) | -22.36 (13.208) | -23.09 (13.890) | -22.49 (14.268)
  Change at Week 44: number analyzed (Participants) | 186 | 178 | 596 | 608
  Change at Week 44 | -22.80 (14.390) | -22.31 (13.062) | -23.19 (14.214) | 23.04 (13.484)
  Change at Week 48: number analyzed (Participants) | 185 | 179 | 599 | 606
  Change at Week 48 | -23.74 (13.685) | -22.56 (13.229) | -23.22 (14.281) | -23.20 (13.008)
  Change at Week 52: number analyzed (Participants) | 190 | 183 | 603 | 617
  Change at Week 52 | -24.09 (13.629) | -23.17 (13.280) | -24.05 (13.930) | -23.61 (13.376)
  Change at Week 76: number analyzed (Participants) | 196 | 185 | 402 | 410
  Change at Week 76 | -27.49 (12.763) | -25.91 (13.537) | -25.98 (14.077) | -24.83 (12.664)
  Change at Week 80: number analyzed (Participants) | 85 | 84 | 174 | 180
  Change at Week 80 | -23.31 (14.840) | -22.67 (12.546) | -23.27 (15.372) | -23.70 (14.755)
  Change at Week 104: number analyzed (Participants) | 280 | 267 | 569 | 573
  Change at Week 104 | -26.85 (13.261) | -26.08 (12.872) | -25.75 (13.931) | -25.60 (13.596)
  Change at Week 128: number analyzed (Participants) | 74 | 74 | 154 | 156
  Change at Week 128 | -24.55 (13.797) | -25.12 (12.102) | -25.06 (15.496) | -26.14 (14.810)
  Change at Week 132: number analyzed (Participants) | 172 | 165 | 347 | 366
  Change at Week 132 | -27.24 (12.671) | -26.62 (13.994) | -26.06 (13.661) | -24.61 (13.391)
  Change at Week 156: number analyzed (Participants) | 238 | 225 | 489 | 503
  Change at Week 156 | -26.53 (14.998) | -26.85 (13.999) | -25.59 (14.641) | -25.60 (13.196)
  Change at Week 180: number analyzed (Participants) | 180 | 168 | 375 | 388
  Change at Week 180 | -27.21 (14.370) | -27.07 (13.969) | -26.95 (13.671) | -25.88 (13.910)
  Change at Week 208: number analyzed (Participants) | 109 | 92 | 197 | 211
  Change at Week 208 | -27.54 (12.054) | -27.06 (15.579) | -27.01 (12.968) | -27.12 (13.008)
  Change at Week 232: number analyzed (Participants) | 34 | 28 | 67 | 69
  Change at Week 232 | -26.61 (13.420) | -26.25 (17.509) | -26.06 (16.858) | -27.23 (14.636)
  Change at Week 260: number analyzed (Participants) | 3 | 2 | 10 | 4
  Change at Week 260 | -34.70 (4.776) | -26.60 (20.789) | -20.73 (11.983) | -19.03 (18.823)

21. Secondary Outcome: Percentage of Participants With Simplified Disease Activity Index Based (SDAI-based) American College of Rheumatology (ACR)/ European League Against Rheumatism (EULAR) Remission Through Week 260
Description: Participant having SDAI-based ACR/EULAR remission at a visit if SDAI score is of <= 3.3. SDAI derived by combining 5 disease assessments: tender joint (28), swollen joint (28) counts, participants global assessment of disease activity using VAS (scale ranges from 0 to 10 [0 =very well to 10 = very poor]), physicians global assessment of disease activity using VAS (scale ranges from 0 to 10 [0=no arthritis to 10=extremely active arthritis]) and CRP. 28 joints evaluated for swelling and tenderness are same set of 28 joints used in DAS28 includes shoulder, elbow, wrist, MCP1, MCP2, MCP3, MCP4, MCP5, PIP1, PIP2, PIP3, PIP4, PIP5 joints of upper right and left extremities and knee joints of lower right and left extremities. Participants were analyzed for efficacy according to assigned treatment groups from the primary studies, regardless of treatments actually received.
Time Frame: Week 2, 4, 6, 8, 12, 16, 18, 20, 24, 28, 32, 36, 40, 44, 48, 52, 76, 80, 104, 128, 132, 156, 180, 208, 232 and 260
Population: as for outcome 17
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo to 50 mg q4w Due to EE/LE/CO | Placebo to 100 mg q2w Due to EE/LE/CO | Sirukumab 50 mg q4w | Sirukumab 100 mg q2w
Number analyzed (Participants) | 305 | 291 | 606 | 618
Percentage of participants
  At Week 2: number analyzed (Participants) | 0 | 0 | 600 | 609
  At Week 2 |  |  | 0.2 | 0.2
  At Week 4: number analyzed (Participants) | 0 | 0 | 596 | 610
  At Week 4 |  |  | 0.8 | 1.1
  At Week 6: number analyzed (Participants) | 0 | 0 | 502 | 522
  At Week 6 |  |  | 1.2 | 2.9
  At Week 8: number analyzed (Participants) | 0 | 0 | 601 | 608
  At Week 8 |  |  | 2.8 | 3.9
  At Week 12: number analyzed (Participants) | 0 | 0 | 598 | 612
  At Week 12 |  |  | 4.5 | 6.4
  At Week 16: number analyzed (Participants) | 0 | 0 | 600 | 611
  At Week 16 |  |  | 5.2 | 8.0
  At Week 18: number analyzed (Participants) | 0 | 0 | 587 | 606
  At Week 18 |  |  | 7.5 | 7.1
  At Week 20: number analyzed (Participants) | 110 | 106 | 600 | 604
  At Week 20 | 0 | 0 | 8.0 | 9.3
  At Week 24: number analyzed (Participants) | 111 | 106 | 603 | 610
  At Week 24 | 1.8 | 1.9 | 9.8 | 10.7
  At Week 28: number analyzed (Participants) | 180 | 172 | 595 | 608
  At Week 28 | 3.9 | 6.4 | 10.4 | 9.2
  At Week 32: number analyzed (Participants) | 177 | 169 | 596 | 607
  At Week 32 | 4.0 | 7.1 | 9.9 | 12.4
  At Week 36: number analyzed (Participants) | 178 | 174 | 596 | 609
  At Week 36 | 4.5 | 7.5 | 11.7 | 13.0
  At Week 40: number analyzed (Participants) | 174 | 172 | 592 | 605
  At Week 40 | 7.5 | 11.0 | 13.7 | 13.7
  At Week 44: number analyzed (Participants) | 184 | 176 | 595 | 605
  At Week 44 | 8.7 | 10.2 | 11.8 | 13.5
  At Week 48: number analyzed (Participants) | 183 | 179 | 591 | 603
  At Week 48 | 8.2 | 12.3 | 14.9 | 12.8
  At Week 52: number analyzed (Participants) | 189 | 181 | 600 | 610
  At Week 52 | 905 | 8.8 | 15.0 | 12.5
  At Week 76: number analyzed (Participants) | 195 | 183 | 399 | 408
  At Week 76 | 16.9 | 13.7 | 16.8 | 14.2
  At Week 80: number analyzed (Participants) | 86 | 83 | 174 | 180
  At Week 80 | 9.3 | 10.8 | 12.6 | 11.1
  At Week 104: number analyzed (Participants) | 279 | 264 | 568 | 571
  At Week 104 | 14.3 | 18.2 | 17.8 | 19.8
  At Week 128: number analyzed (Participants) | 73 | 72 | 155 | 154
  At Week 128 | 8.2 | 15.3 | 16.1 | 13.6
  At Week 132: number analyzed (Participants) | 169 | 165 | 347 | 364
  At Week 132 | 18.3 | 15.8 | 20.5 | 19.0
  At Week 156: number analyzed (Participants) | 235 | 223 | 483 | 499
  At Week 156 | 17.9 | 14.8 | 17.8 | 19.4
  At Week 180: number analyzed (Participants) | 180 | 167 | 374 | 387
  At Week 180 | 18.3 | 20.4 | 22.5 | 24.0
  At Week 208: number analyzed (Participants) | 108 | 92 | 196 | 211
  At Week 208 | 21.3 | 20.7 | 22.4 | 30.3
  At Week 232: number analyzed (Participants) | 27 | 25 | 55 | 57
  At Week 232 | 25.39 | 20.2 | 27.3 | 29.8
  At Week 260: number analyzed (Participants) | 3 | 2 | 9 | 4
  At Week 260 | 33.3 | 50.0 | 55.6 | 0

22. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) Score Through Week 260
Description: The Health Assessment Questionnaire-Disability Index (HAQ-DI) score is an evaluation of the functional status for a participant. The 20-question instrument assesses the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and activities of daily living). Responses in each functional area are scored from 0, indicating no difficulty, to 3, indicating inability to perform a task in that area. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range: 0-3 where 0 = least difficulty and 3 = extreme difficulty. Participants were analyzed for efficacy according to assigned treatment groups from the primary studies, regardless of treatments actually received.
Time Frame: as for outcome 20
Population: Population included all participants who were enrolled in this study. For "Placebo to 50mg" and "Placebo to 100mg" groups, only efficacy data collected after the escape or CO (after Week 18) to sirukumab was planned to be reported, with exception of baseline data. Here 'n' signifies number of participants analyzed at specified time point.
Measure: Mean (Standard Deviation); unit: Units on Scale
Arm/Group | Placebo to 50 mg q4w Due to EE/LE/CO | Placebo to 100 mg q2w Due to EE/LE/CO | Sirukumab 50 mg q4w | Sirukumab 100 mg q2w
Number analyzed (Participants) | 305 | 291 | 606 | 618
Units on Scale
  Change at Week 2: number analyzed (Participants) | 0 | 0 | 603 | 616
  Change at Week 2 |  |  | -0.1136 (0.3455) | -0.1230 (0.3741)
  Change at Week 4: number analyzed (Participants) | 0 | 0 | 602 | 616
  Change at Week 4 |  |  | -0.2307 (0.4173) | -0.2417 (0.4034)
  Change at Week 6: number analyzed (Participants) | 0 | 0 | 511 | 526
  Change at Week 6 |  |  | -0.3112 (0.4944) | -0.3683 (0.4823)
  Change at Week 8: number analyzed (Participants) | 0 | 0 | 602 | 611
  Change at Week 8 |  |  | -0.3499 (0.5077) | -0.3914 (0.5022)
  Change at Week 12: number analyzed (Participants) | 0 | 0 | 601 | 613
  Change at Week 12 |  |  | -0.3866 (0.5421) | -0.4121 (0.5270)
  Change at Week 16: number analyzed (Participants) | 0 | 0 | 606 | 614
  Change at Week 16 |  |  | -0.3991 (0.5611) | -0.4414 (0.5430)
  Change at Week 18: number analyzed (Participants) | 0 | 0 | 602 | 614
  Change at Week 18 |  |  | -0.4365 (0.5476) | -0.4621 (0.5325)
  Change at Week 20: number analyzed (Participants) | 111 | 106 | 602 | 611
  Change at Week 20 | -0.1363 (0.4947) | -0.2005 (0.4987) | -0.4425 (0.5826) | -0.4920 (0.5582)
  Change at Week 24: number analyzed (Participants) | 112 | 106 | 605 | 615
  Change at Week 24 | -0.3192 (0.5279) | -0.3267 (0.4739) | -0.4506 (0.5665) | -0.4876 (0.5622)
  Change at Week 28: number analyzed (Participants) | 180 | 174 | 601 | 612
  Change at Week 28 | -0.3722 (0.5683) | -0.3836 (0.4741) | -0.4736 (0.5696) | -0.4912 (0.5626)
  Change at Week 32: number analyzed (Participants) | 180 | 170 | 601 | 614
  Change at Week 32 | -0.3847 (0.5651) | -0.4015 (0.5532) | -0.4769 (0.5880) | -0.5307 (0.5740)
  Change at Week 36: number analyzed (Participants) | 178 | 174 | 602 | 611
  Change at Week 36 | -0.3862 (0.5474) | -0.4339 (0.5432) | -0.4850 (0.5764) | -0.5176 (0.5688)
  Change at Week 40: number analyzed (Participants) | 177 | 173 | 593 | 613
  Change at Week 40 | -0.4138 (0.5778) | -0.4509 (0.4988) | -0.4850 (0.5894) | -0.5039 (0.5735)
  Change at Week 44: number analyzed (Participants) | 187 | 181 | 597 | 610
  Change at Week 44 | -0.4231 (0.5809) | -0.4461 (0.5206) | -0.4906 (0.6088) | -0.5297 (0.5777)
  Change at Week 48: number analyzed (Participants) | 187 | 179 | 601 | 609
  Change at Week 48 | -0.4392 (0.5911) | -0.4567 (0.5254) | -0.4890 (0.6242) | -0.5470 (0.5942)
  Change at Week 52: number analyzed (Participants) | 191 | 182 | 604 | 618
  Change at Week 52 | -0.4228 (0.5752) | -0.4609 (0.5455) | -0.4946 (0.6021) | -0.5374 (0.5881)
  Change at Week 76: number analyzed (Participants) | 196 | 185 | 402 | 411
  Change at Week 76 | -0.5816 (0.6313) | -0.5351 (0.5605) | -0.5628 (0.6089) | -0.6128 (0.5992)
  Change at Week 80: number analyzed (Participants) | 91 | 87 | 179 | 187
  Change at Week 80 | -0.2074 (0.5333) | -0.3980 (0.5579) | -0.3834 (0.5685) | -0.4211 (0.5626)
  Change at Week 104: number analyzed (Participants) | 282 | 269 | 573 | 579
  Change at Week 104 | -0.4778 (0.6569) | -0.5107 (0.5958) | -0.5153 (0.6094) | -0.5579 (0.5913)
  Change at Week 128: number analyzed (Participants) | 76 | 74 | 157 | 157
  Change at Week 128 | -0.2664 (0.5963) | -0.4476 (0.5263) | -0.3615 (0.6227) | -0.4506 (0.5527)
  Change at Week 132: number analyzed (Participants) | 178 | 169 | 362 | 375
  Change at Week 132 | -0.4831 (0.6979) | -0.4815 (0.6656) | -0.5045 (0.6542) | -0.5310 (0.6240)
  Change at Week 156: number analyzed (Participants) | 243 | 231 | 503 | 505
  Change at Week 156 | -0.4614 (0.6610) | -0.4984 (0.6520) | -0.4719 (0.6604) | -0.4998 (0.6109)
  Change at Week 180: number analyzed (Participants) | 187 | 276 | 384 | 393
  Change at Week 180 | -0.4505 (0.7024) | -0.4957 (0.5969) | -0.5072 (0.6492) | -0.5258 (0.6167)
  Change at Week 208: number analyzed (Participants) | 109 | 94 | 201 | 217
  Change at Week 208 | -0.4622 (0.6898) | -0.4973 (0.6032) | -0.5031 (0.6701) | -0.5588 (0.6023)
  Change at Week 232: number analyzed (Participants) | 34 | 29 | 67 | 69
  Change at Week 232 | -0.4191 (0.7410) | -0.4655 (0.6477) | -0.5877 (0.8312) | -0.6069 (0.6262)
  Change at Week 260: number analyzed (Participants) | 3 | 2 | 9 | 3
  Change at Week 260 | -0.5417 (0.8323) | -0.3750 (1.0607) | -0.2083 (0.6702) | -0.5000 (0.4507)

23. Secondary Outcome: Percentage of Participants With Health Assessment Questionnaire-Disability Index (HAQ-DI) Response Through Week 260
Description: HAQ-DI response was defined as change of less than -0.22 from baseline in HAQ-DI score. The HAQ-DI score is an evaluation of the functional status for a participant. The 20-question instrument assesses the degree of difficulty a person has in accomplishing tasks in 8 functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and activities of daily living). Responses in each functional area are scored from 0, indicating no difficulty, to 3, indicating inability to perform a task in that area. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0-3 where 0 = least difficulty and 3 = extreme difficulty. Participants were analyzed for efficacy according to assigned treatment groups from the primary studies, regardless of treatments actually received.
Time Frame: Week 2, 4, 6, 8, 12, 16, 18, 20, 24, 28, 32, 36, 40, 44, 48, 52, 76, 80, 104, 128, 132, 156, 180, 208, 232 and 260
Population: as for outcome 17
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo to 50 mg q4w Due to EE/LE/CO | Placebo to 100 mg q2w Due to EE/LE/CO | Sirukumab 50 mg q4w | Sirukumab 100 mg q2w
Number analyzed (Participants) | 305 | 291 | 606 | 618
Percentage of participants
  At Week 2: number analyzed (Participants) | 0 | 0 | 603 | 616
  At Week 2 |  |  | 36.3 | 36.4
  At Week 4: number analyzed (Participants) | 0 | 0 | 602 | 616
  At Week 4 |  |  | 48.3 | 51.3
  At Week 6: number analyzed (Participants) | 0 | 0 | 511 | 526
  At Week 6 |  |  | 56.4 | 57.6
  At Week 8: number analyzed (Participants) | 0 | 0 | 602 | 611
  At Week 8 |  |  | 58.0 | 62.5
  At Week 12: number analyzed (Participants) | 0 | 0 | 601 | 613
  At Week 12 |  |  | 60.4 | 62.3
  At Week 16: number analyzed (Participants) | 0 | 0 | 602 | 614
  At Week 16 |  |  | 62.0 | 63.2
  At Week 18: number analyzed (Participants) | 0 | 0 | 602 | 614
  At Week 18 |  |  | 63.0 | 66.0
  At Week 20: number analyzed (Participants) | 111 | 106 | 602 | 611
  At Week 20 | 40.5 | 45.3 | 64.0 | 67.1
  At Week 24: number analyzed (Participants) | 112 | 106 | 605 | 615
  At Week 24 | 54.5 | 54.7 | 64.3 | 67.0
  At Week 28: number analyzed (Participants) | 180 | 174 | 601 | 612
  At Week 28 | 58.3 | 61.5 | 66.7 | 66.8
  At Week 32: number analyzed (Participants) | 180 | 170 | 601 | 614
  At Week 32 | 59.4 | 59.4 | 65.2 | 68.1
  At Week 36: number analyzed (Participants) | 178 | 174 | 602 | 611
  At Week 36 | 61.2 | 64.9 | 67.1 | 67.9
  At Week 40: number analyzed (Participants) | 177 | 173 | 593 | 613
  At Week 40 | 61.0 | 67.1 | 65.4 | 66.6
  At Week 44: number analyzed (Participants) | 187 | 181 | 597 | 610
  At Week 44 | 62.6 | 65.2 | 65.8 | 67.9
  At Week 48: number analyzed (Participants) | 187 | 179 | 601 | 609
  At Week 48 | 61.5 | 65.9 | 65.6 | 70.1
  At Week 52: number analyzed (Participants) | 191 | 182 | 604 | 618
  At Week 52 | 60.7 | 65.9 | 65.6 | 68.9
  At Week 76: number analyzed (Participants) | 196 | 185 | 598 | 411
  At Week 76 | 70.4 | 69.2 | 68.4 | 73.7
  At Week 80: number analyzed (Participants) | 91 | 87 | 179 | 187
  At Week 80 | 40.7 | 58.6 | 58.1 | 62.0
  At Week 104: number analyzed (Participants) | 282 | 269 | 573 | 579
  At Week 104 | 64.2 | 68.4 | 66.1 | 68.0
  At Week 128: number analyzed (Participants) | 76 | 74 | 157 | 157
  At Week 128 | 51.3 | 64.9 | 54.8 | 61.1
  At Week 132: number analyzed (Participants) | 178 | 169 | 362 | 375
  At Week 132 | 65.2 | 63.3 | 66.3 | 69.9
  At Week 156: number analyzed (Participants) | 243 | 231 | 503 | 505
  At Week 156 | 62.6 | 64.5 | 65.0 | 66.9
  At Week 180: number analyzed (Participants) | 187 | 176 | 384 | 393
  At Week 180 | 61.0 | 69.3 | 66.4 | 72.3
  At Week 208: number analyzed (Participants) | 109 | 94 | 201 | 217
  At Week 208 | 65.1 | 69.1 | 71.1 | 72.4
  At Week 232: number analyzed (Participants) | 34 | 29 | 67 | 69
  At Week 232 | 67.6 | 69.0 | 65.7 | 72.5
  At Week 260: number analyzed (Participants) | 3 | 2 | 9 | 3
  At Week 260 | 66.7 | 50.0 | 44.4 | 66.7

ADVERSE EVENTS:
Time Frame: Baseline of this LTE study through up to 4.3 years
Description: Population included all participants who were enrolled in this study. 1 participant who mistakenly took sirukumab 100mg, when was originally assigned to sirukumab 50mg, was analyzed under the sirukumab 100mg group for all safety analyses. In treatment group 'Placebo to 100 mg q2w Due to EE/LE/CO', 6 deaths happened during the CNTO136ARA3004 study. One additional death was reported in this group after the participant was discontinued from the study.
Arm/Group | Placebo to 50 mg q4w Due to EE/LE/CO | Placebo to 100 mg q2w Due to EE/LE/CO | Sirukumab 50 mg q4w | Sirukumab 100 mg q2w
All-Cause Mortality (participants affected / at risk) | 5/305 | 7/291 | 13/605 | 8/619
Serious Adverse Events (participants affected / at risk) | 65/305 | 81/291 | 160/605 | 143/619
Other Adverse Events (participants affected / at risk) | 139/305 | 135/291 | 268/605 | 281/619
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo to 50 mg q4w Due to EE/LE/CO (N=305) | Placebo to 100 mg q2w Due to EE/LE/CO (N=291) | Sirukumab 50 mg q4w (N=605) | Sirukumab 100 mg q2w (N=619)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Hypochromic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 3 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Acute left ventricular failure (Cardiac disorders) | 0 | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 3 | 3
Angina pectoris (Cardiac disorders) | 0 | 0 | 2 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 3 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 2 | 6
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac tamponade (Cardiac disorders) | 1 | 0 | 0 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0 | 1 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1 | 0
Coronary artery insufficiency (Cardiac disorders) | 0 | 0 | 1 | 0
Hypertensive heart disease (Cardiac disorders) | 0 | 0 | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 0 | 0
Pericarditis (Cardiac disorders) | 1 | 0 | 0 | 0
Sinus node dysfunction (Cardiac disorders) | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Hydrocele (Congenital, familial and genetic disorders) | 1 | 0 | 1 | 0
Inner ear disorder (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Meniere's disease (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1 | 0
Blindness (Eye disorders) | 0 | 0 | 0 | 1
Cataract (Eye disorders) | 1 | 1 | 3 | 0
Corneal perforation (Eye disorders) | 0 | 0 | 0 | 1
Keratitis (Eye disorders) | 0 | 0 | 1 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 1 | 0
Scleritis (Eye disorders) | 0 | 0 | 1 | 0
Ulcerative keratitis (Eye disorders) | 0 | 1 | 0 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 2 | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diverticular perforation (Gastrointestinal disorders) | 1 | 1 | 1 | 3
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastric volvulus (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Gastrointestinal angiodysplasia haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Haemorrhoids thrombosed (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 2 | 0 | 1
Mesenteric vein thrombosis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pancreatic cyst (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Chest pain (General disorders) | 1 | 1 | 1 | 0
Death (General disorders) | 1 | 0 | 1 | 0
Implant site haematoma (General disorders) | 0 | 0 | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 1
Peripheral swelling (General disorders) | 0 | 0 | 0 | 1
Soft tissue inflammation (General disorders) | 0 | 1 | 0 | 0
Sudden cardiac death (General disorders) | 0 | 0 | 1 | 1
Biliary colic (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 2 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 2 | 1 | 1
Sphincter of Oddi dysfunction (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Abscess (Infections and infestations) | 0 | 0 | 1 | 0
Abscess intestinal (Infections and infestations) | 0 | 0 | 0 | 1
Abscess limb (Infections and infestations) | 2 | 1 | 0 | 1
Anal abscess (Infections and infestations) | 0 | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 2 | 1
Arthritis bacterial (Infections and infestations) | 1 | 1 | 2 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0
Bacterial pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 0
Beta haemolytic streptococcal infection (Infections and infestations) | 0 | 0 | 1 | 0
Breast abscess (Infections and infestations) | 0 | 0 | 1 | 0
Breast cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 1
Bursitis infective staphylococcal (Infections and infestations) | 1 | 0 | 0 | 2
Cellulitis (Infections and infestations) | 3 | 4 | 12 | 10
Colonic abscess (Infections and infestations) | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 2 | 0
Dermatitis infected (Infections and infestations) | 0 | 0 | 1 | 0
Device related infection (Infections and infestations) | 1 | 1 | 0 | 1
Diverticulitis (Infections and infestations) | 2 | 1 | 1 | 2
Erysipelas (Infections and infestations) | 0 | 0 | 4 | 5
Extradural abscess (Infections and infestations) | 0 | 0 | 1 | 0
Gangrene (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis salmonella (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 1
Haematoma infection (Infections and infestations) | 0 | 1 | 0 | 0
Hepatitis E (Infections and infestations) | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 1 | 0 | 1
Herpes zoster disseminated (Infections and infestations) | 0 | 0 | 1 | 0
Infected seroma (Infections and infestations) | 0 | 0 | 0 | 1
Infected skin ulcer (Infections and infestations) | 1 | 0 | 0 | 0
Infectious pleural effusion (Infections and infestations) | 0 | 0 | 1 | 0
Infective tenosynovitis (Infections and infestations) | 0 | 0 | 1 | 0
Intervertebral discitis (Infections and infestations) | 0 | 0 | 1 | 0
Klebsiella infection (Infections and infestations) | 0 | 1 | 0 | 0
Localised infection (Infections and infestations) | 0 | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 2 | 0 | 1 | 0
Mastitis (Infections and infestations) | 0 | 0 | 0 | 1
Medical device site joint infection (Infections and infestations) | 0 | 0 | 0 | 1
Meningitis pneumococcal (Infections and infestations) | 0 | 0 | 0 | 1
Necrotising fasciitis (Infections and infestations) | 1 | 0 | 2 | 0
Ophthalmic herpes zoster (Infections and infestations) | 0 | 0 | 1 | 1
Osteomyelitis (Infections and infestations) | 2 | 1 | 2 | 3
Peritonitis (Infections and infestations) | 0 | 1 | 1 | 1
Pilonidal cyst (Infections and infestations) | 0 | 0 | 0 | 1
Pneumococcal sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 4 | 8 | 9 | 19
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 1 | 1
Pneumonia pneumococcal (Infections and infestations) | 1 | 1 | 0 | 0
Pneumonia viral (Infections and infestations) | 0 | 1 | 0 | 0
Post procedural infection (Infections and infestations) | 0 | 0 | 1 | 1
Postoperative wound infection (Infections and infestations) | 0 | 1 | 1 | 0
Psoas abscess (Infections and infestations) | 0 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 1 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 2 | 0
Pyomyositis (Infections and infestations) | 1 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 1 | 6 | 3 | 5
Septic shock (Infections and infestations) | 1 | 3 | 0 | 2
Soft tissue infection (Infections and infestations) | 0 | 0 | 0 | 1
Spinal cord infection (Infections and infestations) | 0 | 0 | 0 | 1
Staphylococcal abscess (Infections and infestations) | 0 | 0 | 0 | 2
Staphylococcal infection (Infections and infestations) | 0 | 1 | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 1 | 0
Staphylococcal skin infection (Infections and infestations) | 0 | 0 | 0 | 1
Streptococcal abscess (Infections and infestations) | 0 | 0 | 0 | 1
Streptococcal endocarditis (Infections and infestations) | 0 | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 1
Tuberculosis (Infections and infestations) | 1 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 2 | 2
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 1
Vulval abscess (Infections and infestations) | 0 | 0 | 0 | 1
Wound infection (Infections and infestations) | 0 | 0 | 1 | 0
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Comminuted fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Dislocation of vertebra (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 | 1 | 2 | 1
Femur fracture (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 1
Fractured sacrum (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 2 | 2 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Muscle injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Post procedural fistula (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Postoperative thrombosis (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Skin injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 2 | 0
Splenic rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Synovial rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Wound necrosis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Transaminases increased (Investigations) | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 1
Atlantoaxial instability (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0
Finger deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3 | 0
Mixed connective tissue disease (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 9 | 3 | 9
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 6 | 5
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Acute promyelocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Benign ovarian tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 3
Central nervous system lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Inflammatory pseudotumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Monoclonal gammopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Renal cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Schwannoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Squamous cell carcinoma of pharynx (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Vaginal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 0 | 1
Cerebellar infarction (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebral artery embolism (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebral haematoma (Nervous system disorders) | 0 | 0 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 4 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 1 | 1 | 3
Cubital tunnel syndrome (Nervous system disorders) | 0 | 0 | 0 | 1
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 0 | 1 | 0
Facial paresis (Nervous system disorders) | 1 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 1 | 0
Hypertensive encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1
IIIrd nerve paralysis (Nervous system disorders) | 0 | 0 | 0 | 1
Intracranial mass (Nervous system disorders) | 0 | 1 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0 | 0
Lumbar radiculopathy (Nervous system disorders) | 0 | 0 | 1 | 0
Mononeuropathy multiplex (Nervous system disorders) | 1 | 0 | 0 | 0
Myxoedema coma (Nervous system disorders) | 0 | 0 | 1 | 0
Spondylitic myelopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 2 | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 1 | 1
Ulnar tunnel syndrome (Nervous system disorders) | 1 | 0 | 0 | 0
Device dislocation (Product Issues) | 0 | 1 | 2 | 0
Device loosening (Product Issues) | 0 | 0 | 0 | 1
Acute psychosis (Psychiatric disorders) | 0 | 0 | 1 | 0
Alcohol abuse (Psychiatric disorders) | 0 | 1 | 0 | 0
Conversion disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 3 | 0
Depression suicidal (Psychiatric disorders) | 0 | 0 | 1 | 0
Disorientation (Psychiatric disorders) | 0 | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 1
Persistent depressive disorder (Psychiatric disorders) | 0 | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 2 | 5
Calculus urethral (Renal and urinary disorders) | 0 | 0 | 1 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 1 | 0 | 0
Cystitis interstitial (Renal and urinary disorders) | 0 | 0 | 0 | 1
Glomerulonephritis (Renal and urinary disorders) | 0 | 0 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 2 | 0
IgA nephropathy (Renal and urinary disorders) | 0 | 0 | 0 | 1
Incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1
Lupus nephritis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 3 | 2
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal haematoma (Renal and urinary disorders) | 1 | 0 | 0 | 0
Stag horn calculus (Renal and urinary disorders) | 0 | 0 | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 0 | 1 | 3 | 0
Cervical polyp (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Endometriosis (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Genital haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Pelvic prolapse (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Uterine polyp (Reproductive system and breast disorders) | 0 | 0 | 0 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 3
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 2
Diaphragmatic disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 2
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hypersensitivity vasculitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 5 | 1
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Aortic aneurysm (Vascular disorders) | 0 | 0 | 1 | 0
Aortic dissection (Vascular disorders) | 1 | 1 | 0 | 0
Aortic stenosis (Vascular disorders) | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 1 | 2 | 2
Hypertension (Vascular disorders) | 0 | 1 | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 0 | 3 | 0
Malignant hypertension (Vascular disorders) | 0 | 0 | 1 | 0
Penetrating aortic ulcer (Vascular disorders) | 0 | 0 | 1 | 0
Peripheral vascular disorder (Vascular disorders) | 0 | 1 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 1 | 0 | 0
Varicose vein (Vascular disorders) | 1 | 0 | 0 | 0
Vasculitis (Vascular disorders) | 0 | 0 | 0 | 1
Vasculitis necrotising (Vascular disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo to 50 mg q4w Due to EE/LE/CO (N=305) | Placebo to 100 mg q2w Due to EE/LE/CO (N=291) | Sirukumab 50 mg q4w (N=605) | Sirukumab 100 mg q2w (N=619)
Leukopenia (Blood and lymphatic system disorders) | 5 | 14 | 23 | 33
Injection site erythema (General disorders) | 10 | 17 | 16 | 26
Bronchitis (Infections and infestations) | 29 | 20 | 32 | 41
Upper respiratory tract infection (Infections and infestations) | 30 | 35 | 52 | 62
Urinary tract infection (Infections and infestations) | 11 | 15 | 24 | 17
Viral upper respiratory tract infection (Infections and infestations) | 37 | 36 | 73 | 80
Alanine aminotransferase increased (Investigations) | 27 | 29 | 35 | 47
Aspartate aminotransferase increased (Investigations) | 16 | 18 | 22 | 35
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 35 | 30 | 80 | 65
Hypertension (Vascular disorders) | 14 | 14 | 31 | 31

LIMITATIONS AND CAVEATS:
Due to early study termination, full intended length of observation and amount of safety, efficacy data collected for participants receiving sirukumab was not achieved and only statistical analysis plan dedicated to safety data(Week 28) was created.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2016-10-06): https://cdn.clinicaltrials.gov/large-docs/09/NCT01856309/Prot_000.pdf
  • Statistical Analysis Plan (2019-04-09): https://cdn.clinicaltrials.gov/large-docs/09/NCT01856309/SAP_001.pdf